CLINICAL TRIAL: NCT05039736
Title: A Phase II Study to Evaluate the Effects of Sequential Therapy With the Anti c-MET/VEGFR Tyrosine Kinase Inhibitor (TKI), Cabozantinib, Followed by an Anti-PD-1 Antibody (Nivolumab) in Patients With Advanced HCC Who Progressed on First-line Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: 0 participants accrued
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0680; NCI-2021-09178 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2021-09-01; First posted 2021-09-10 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — cabozantinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- cabozantinib (Experimental): cabozantinib by mouth every day for 6 weeks
  Interventions: Drug: Cabozantinib
- nivolumab (Experimental): nivolumab by vein every 4 weeks for up to 2 years
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Cabozantinib — Given by PO
  Other Names: XL-184; XL184
  Arms: cabozantinib
Drug: Nivolumab — Given by IV
  Other Names: BMS-936558; Opdivo
  Arms: nivolumab

SUMMARY:
The purpose of this clinical research study is to learn about the safety and effectiveness of cabozantinib and nivolumab in people with hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Primary objective is to evaluate overall response rate

Secondary objectives are to evaluate progression-free survival and overall survival

Exploratory endpoints

To explore the association between c-MET, PD-1/PD-L1 (and PD-L2) expression by immunohistochemistry, RNA seq genomic profiling and antitumor efficacy of nivolumab

+ cabozantinib based on RECIST 1.1 To evaluate correlation between fibrosis stage by histology, by magnetic resonance elastography (MRE) imaging and by IGF1 scores To evaluate baseline and longitudinal changes of blood and tumor markers such as TNFα, pSTAT3, and EGFR, immune cell density including frequency of PD-1 + 4-1BB + CD8+ T cells, pro-inflammatory cytokines, and hepatic fibrosis markers (APRI, FIB-4, hyaluronic acid, FibroTest [FibroSure], nonalcoholic fatty-liver disease fibrosis score, enhanced liver fibrosis [ELF]) test as biomarkers of response to therapy To evaluate candidate serum and tissue biomarkers to predict response to cabozantinib (e.g. Kallikrein 5, KLK-7, MCP-1, LAP/TGF-β1, Galectin-3) and nivolumab (e.g. angiogenin, Endostatin, PGI, PAI-1, Cystatin-B, CD8 T cell frequency and Ki67) To evaluate the predictive value of dynamic changes in fibrosis stage (defined by a minimum 2-point improvement in fibrosis grade 0-4 per MRE) and in IGF-1 blood scores

ELIGIBILITY:
Inclusion Criteria

* Is willing and able to provide written informed consent for the trial. Consent for Future Biomedical Research is optional-the subject may participate in the main trial without participating in Future Biomedical Research.
* Has a histologically or cytologically confirmed diagnosis of HCC (fibrolamellar and mixed hepatocellular/cholangiocarcinoma subtypes are not eligible) confirmed by a pathologist at
* Has Barcelona Clinic Liver Cancer (BCLC) Stage-C disease or BCLC Stage-B disease not amenable to locoregional therapy or refractory to locoregional therapy and not amenable to a curative treatment approach (see Appendix 12.8).
* Has a Child-Pugh A liver score within 7 days of first dose of study drug.
* Has documented objective radiographic progression after at least one line of therapy with sorafenib, lenvatinib, bevacizumab, regorafenib, ramucirumab, and immune checkpoint inhibitors including nivolumab, atezolizumab, pembrolizumab, ipilimumab, avelumab, durvalumab, and tremelimumab, or had intolerance to sorafenib, lenvatinib, regorafenib, bevacizumab, or ramucirumab.
* Has measurable disease based on RECIST 1.1 as confirmed by the MD Anderson radiologist.

Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.

* Patients who have chronic, untreated hepatitis C virus (HCV) are allowed. Has recovered to baseline or ≤ Grade 1 CTCAE v5.0 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
* Has a performance status of 0 or 1 using the Eastern Cooperative Oncology Group performance status scale within 7 days of first dose of study drug.
* Has adequate organ and marrow function, based upon meeting all of the following laboratory criteria within 7 days before first dose of study treatment
* Has a negative urine or serum pregnancy test (if female) within 72 hours prior to receiving the first dose of study medication (Cycle 1, Day 1) (female subjects of childbearing potential). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception during the course of the study and for 1 year after the last dose of study treatment.

Acceptable methods of contraception are as follows:

* Single method (one of the following is acceptable):

  * intrauterine device (IUD)
  * vasectomy of a female subject's male partner
  * contraceptive rod implanted into the skin
* Combination method (requires use of two of the following):

  * diaphragm with spermicide (cannot be used in conjunction with cervical cap/spermicide) cervical cap with spermicide (nulliparous women only)
  * contraceptive sponge (nulliparous women only)
  * male condom or female condom (cannot be used together)
  * hormonal contraceptive: oral contraceptive pill (estrogen/progestin pill or progestin- only pill), contraceptive skin patch, vaginal contraceptive ring, or subcutaneous contraceptive injection
* Abstinence is acceptable if this is the usual lifestyle and preferred contraception method for the subject.

  * Female subjects of childbearing potential must not be pregnant at screening. Females of childbearing potential are defined as premenopausal females capable of becoming pregnant (ie, females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti-estrogens, low body weight, ovarian suppression or other reasons.
  * Among patients deemed to be eligible, those who were treated with anti-viral medications and recovered from COVID-19 must undergo a two-week washout period before initiation of cabozantinib. Asymptomatic patients who tested positive are required to remain asymptomatic for two weeks before starting cabozantinib.
  * Must have biopsy-eligible lesions for mandatory biopsies.

Exclusion Criteria

* Received prior treatment with cabozantinib.
* Has participated (or is currently participating) in a study of an investigational agent and received (or is receiving) study therapy, herbal/complementary oral or IV medicine including cytotoxic, biologic, or other systemic anticancer therapy, or used (is using) an investigation device, other than sorafenib, lenvatinib, bevacizumab, regorafenib, ramucirumab, and immune checkpoint inhibitors including nivolumab, atezolizumab, pembrolizumab, ipilimumab, avelumab, durvalumab, and tremelimumab, within 4 weeks of the first dose of treatment. Subjects must also have recovered from associated therapy (i.e., to Grade ≤1 or baseline) and from adverse events due to any prior therapy.
* Has developed grade 3 or higher adverse events from prior immune checkpoint inhibitors including nivolumab, atezolizumab, pembrolizumab, ipilimumab, avelumab, durvalumab, and tremelimumab and could not continue the treatment are excluded..
* Had esophageal or gastric variceal bleeding within the last 6 months. All subjects will be screened for esophageal varices, unless such screening has been performed in the past 12 months before first dose of treatment. If varices are present, they should be treated according to institutional standards before starting study treatment.
* Has an ALT >5x upper limit of normal (ULN) on Day 1 of study treatment.
* Has a total bilirubin >2.0 mg/dL on Day 1 of study treatment.
* Has clinically apparent ascites or encephalopathy, or untreated varices. Must have undergone an upper endoscopy within 3 months from trial and treated per institutional guidelines for esophageal varices to be eligible.
* Has portal vein HCC invasion at the main portal branch (Vp4) or inferior vena cava, or has cardiac involvement of HCC based on imaging.
* Had encephalopathy in the last 6 months. Subjects on rifaximin or lactulose to control their encephalopathy are not allowed.
* Had a solid organ or hematologic transplant.
* Received radiation therapy for bone metastasis within 2 weeks, and any other radiation therapy within 4 weeks, before first dose of study treatment. Received systemic treatment with radionuclides within 6 weeks before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* Has active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.

The use of physiologic doses of corticosteroids may be approved after consultation with BMS/Exelixis or IND Office. -Has received locoregional therapy to liver (TACE, TAE, radiation, radioembolization, or ablation) or surgery to liver or other site within 6 weeks prior to the first dose of study drug.

Minor surgery (e.g., simple excision, tooth extraction) must have occurred at least 7 days prior to the first dose of study treatment (Cycle 1, Day 1). Subjects must have recovered adequately (i.e., Grade ≤1 or baseline) from the toxicity and/or complications from any intervention prior to starting therapy.

* Has a diagnosed additional malignancy within 5 years prior to first dose of study treatment with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or curatively resected in situ cervical and/or breast cancers.
* Has radiographically detectable (even if asymptomatic and/or previously treated) central nervous system metastases and/or carcinomatous meningitis as assessed by local site investigator and radiology review.
* Has a known history of, or any evidence of, interstitial lung disease or active non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy (including dialysis), or laboratory abnormality that might confound the results of the trial or might interfere with the subject's participation for the full duration of the trial, in the opinion of the treating investigator. Or it is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 1 year after the last dose of trial treatment.
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has untreated active HBV. Note: To qualify for enrollment, antiviral therapy for HBV must be given for at least 3 months prior to first dose of study drug, and HBV viral load must be less than 100 IU/mL prior to first dose of study drug. Those on active HBV therapy with viral loads under 100 IU/mL should stay on the same therapy throughout study treatment. Those subjects who are anti-HBc (+) and negative for HBsAg, Anti-HBs, and HBV viral load do not require HBV prophylaxis, but need close monitoring for reactivation as described in Section 5.6.2.
* Has hepatitis C and has received therapy for HCV <4 weeks from the start of current trial therapy. Note: Those with untreated HCV and those who completed HCV therapy ≥4 weeks of study treatment start are eligible.
* Has dual infection with HBV/HCV or other hepatitis combinations at study entry.
* Has received a live or live-attenuated vaccine (eg, intranasal influenza vaccines or FluMist®) within 30 days of planned start of study therapy (Cycle 1, Day 1). Killed virus vaccines used for seasonal influenza vaccines for injection are allowed.
* Is receiving concomitant anticoagulation with oral anticoagulants (eg, warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (eg, clopidogrel).

Allowed anticoagulants are the following:

1. Low-dose aspirin for cardioprotection (per local applicable guidelines) is permitted.
2. Low-dose low molecular-weight heparins (LMWH) are permitted.
3. Anticoagulation with therapeutic doses of LMWH is allowed in subjects without known brain metastases who are on a stable dose of LMWH for at least 2 weeks before first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.

   * Has prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) ≥ 1.5 × the laboratory ULN within 7 days before the first dose of study treatment
   * Has uncontrolled, significant, intercurrent or recent illness including, but not limited to, the following conditions:

a. Cardiovascular disorders: i. Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias. ii. Uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment. iii. Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (eg, deep venous thrombosis, pulmonary embolism) within 6 months before first dose. b. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation: i. Tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (eg, Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction. ii. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose. c. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose. d. Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation. e. Lesions invading or encasing any major blood vessels. f. Other clinically significant disorders that would preclude safe study participation.

i. Serious non-healing wound/ulcer/bone fracture. ii. Uncompensated/symptomatic hypothyroidism. iii. Moderate to severe hepatic impairment (Child-Pugh B or -C).

* Had major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 8 weeks before first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before first dose and from minor surgery (eg, simple excision, tooth extraction) at least 10 days before first dose. Subjects with clinically relevant, ongoing complications from prior surgery are not eligible.
* Has a corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 28 days before first dose of study treatment (https://www.ahajournals.org/doi/10.1161/JAHA.116.003264). Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 minutes must be performed within 30 minutes after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.
* Is unable to swallow tablets.
* Has a previously identified allergy or hypersensitivity to components of the study treatment formulations.
* Has active severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-24 (Estimated); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
To evaluate overall response rate | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sunyoung Lee, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org